CLINICAL TRIAL: NCT07359638
Title: The Effects of a Mandibular Oral Repositioning Device on Sleep Quality, Heart Rate Variability, & SpO2
Brief Title: Impact of a Mandibular Oral Repositioning Device on Sleep Quality, Heart Rate Variability, & SpO2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Sport Institute Alberta (Unknown); PX3 (Unknown)
Responsible Party: Principal Investigator, Christian Clermont, Adjunct Assistant Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: REB25-1741
Record Dates: First submitted 2025-12-22; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sleep
Keywords: mandibular oral appliance; sleep quality; heart rate variability; oxygen saturation; airway patency
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- px3 (Experimental): The PX3™ Mandibular Oral Repositioning Appliance is designed to advance and stabilize the lower jaw, optimizing airway openness and physiological efficiency. The device functions similarly to the airway-opening maneuver used in cardiopulmonary resuscitation, slightly bringing the mandible forward to facilitate airflow. Each PX3™ appliance is custom-fitted to align and lock opposing teeth, stabilizing the jaw during sleep or high-stress activities.
  PX3™ designs are based on three physical principles:
  (i) Poiseuille's Law: Increasing airway volume increases oxygen intake. (ii) Gas Exchange Law: Optimized oxygen and carbon dioxide exchange enhances physiological function.
  (iii) Conservation of Energy Law: Greater oxygen availability improves mechanical efficiency.
  Interventions: Device: Mandibular Oral Repositioning Appliance
- Placebo Device (Placebo Comparator): The Placebo Device is a splint in centric occlusion with no mandibular advancement. The PX3™ Device advances the mandible 50-70% of maximum protrusion to improve alignment.
  Interventions: Device: Mandibular Oral Repositioning Appliance

INTERVENTIONS:
Device: Mandibular Oral Repositioning Appliance — The PX3™ Mandibular Oral Repositioning Appliance is designed to advance and stabilize the lower jaw, optimizing airway openness and physiological efficiency. The device functions similarly to the airway-opening maneuver used in cardiopulmonary resuscitation, slightly bringing the mandible forward to facilitate airflow. Each PX3™ appliance is custom-fitted to align and lock opposing teeth, stabilizing the jaw during sleep or high-stress activities.
  PX3™ designs are based on three physical principles:
  (i) Poiseuille's Law: Increasing airway volume increases oxygen intake. (ii) Gas Exchange Law: Optimized oxygen and carbon dioxide exchange enhances physiological function.
  (iii) Conservation of Energy Law: Greater oxygen availability improves mechanical efficiency.

SUMMARY:
Fatigue, poor sleep quality, and reduced physiological recovery are common even among otherwise healthy adults. Subtle factors such as jaw position during sleep and breathing efficiency may contribute to these issues. The mandible (lower jaw) is suspended by muscles and ligaments rather than fixed joints, making it susceptible to small positional changes during sleep. Even mild misalignment of the lower jaw can reduce airway space, alter breathing mechanics, and disrupt sleep architecture, which may in turn affect autonomic regulation and recovery.

This study will evaluate whether a custom mandibular oral repositioning appliance (px3™) improves sleep quality and recovery-related physiological measures compared with a placebo oral device. The px3™ device gently advances the lower jaw during sleep, which may help maintain airway openness and support more stable breathing. The placebo device is custom-fitted but holds the jaw in a neutral position without mandibular advancement, allowing for controlled comparison of device effects.

Using a randomized crossover design, each participant will wear both the px3™ device and the placebo device during separate intervention phases, allowing participants to serve as their own control. The study will take place over approximately 12 weeks and includes baseline monitoring without any oral appliance, two intervention phases, a washout period between conditions, and a short follow-up period.

Participants will undergo non-invasive digital dental scans to fabricate two custom oral devices. Sleep, heart rate variability (HRV), and blood oxygen saturation (SpO₂) will be continuously monitored using a wrist-worn wearable device throughout the study, except during bathing or charging. Participants will also complete brief questionnaires and sleep logs to report comfort, adherence, perceived effects, and factors that may influence sleep (e.g., illness, travel, or alcohol use).

The primary outcomes of interest are changes in sleep stage distribution (including deep, light, and REM sleep), HRV, and SpO₂ when using the PX3™ device compared with the placebo device. Secondary outcomes include participant comfort, adherence, and user experience. The findings from this study will help determine whether mandibular oral repositioning may support sleep quality and physiological recovery in healthy adults.

DETAILED DESCRIPTION:
1. Background and Rationale

   Fatigue, stress, and burnout are increasingly prevalent among healthy, high-performance individuals. Two often-overlooked contributors are jaw misalignment (malocclusion) and over-breathing, both of which can impair respiratory efficiency, sleep quality, and physiological recovery.

   The mandible is unique in the human body, suspended by muscles and ligaments rather than fixed joints. This provides a wide range of motion but makes it susceptible to misalignment during activity or sleep. Even mild malocclusion can compromise airway patency, neuromuscular coordination, and craniofacial balance. Consequences may include reduced respiratory efficiency, increased fatigue, impaired concentration, and elevated injury risk. Secondary issues from mouth-breathing and over-breathing - such as poor oxygen-carbon dioxide balance and disrupted sleep - further contribute to fatigue and suboptimal performance.

   The PX3™ Mandibular Oral Repositioning Appliance is designed to advance and stabilize the lower jaw, optimizing airway openness and physiological efficiency. The device functions similarly to the airway-opening maneuver used in cardiopulmonary resuscitation, slightly bringing the mandible forward to facilitate airflow. Each PX3™ appliance is custom-fitted to align and lock opposing teeth, stabilizing the jaw during sleep or high-stress activities.

   PX3™ designs are based on three physical principles:

   (i) Poiseuille's Law: Increasing airway volume increases oxygen intake. (ii) Gas Exchange Law: Optimized oxygen and carbon dioxide exchange enhances physiological function.

   (iii) Conservation of Energy Law: Greater oxygen availability improves mechanical efficiency.

   Preliminary PX3™ testing has shown positive trends in airway efficiency, strength, balance, and endurance. In a study by Zupan et al. (2018), 25 participants demonstrated significantly faster 1.5-mile run times, greater anaerobic endurance, and higher leg-press strength when using the PX3™ device compared with a standard mouthguard or no mouthpiece. Nevertheless, the effects of this intervention on sleep quality and heart rate variability (HRV) - markers of recovery and autonomic balance - have not been evaluated in a controlled research setting.
2. Research Question & Objectives:

   Research Question: Does the PX3™ Mandibular Oral Repositioning Appliance improve sleep quality, heart rate variability, and blood oxygen saturation (SpO2) in healthy adults?

   Objectives:

   (i) To determine whether wearing the PX3™ appliance during sleep changes sleep stage distribution (deep, light, REM, awake), HRV, and SpO2 compared with a placebo device.

   (ii) To evaluate participant experience, comfort, and adherence.
3. Methods:

Study Design:

A randomized crossover design will compare the effects of the PX3™ device versus a placebo oral appliance. Each participant will complete baseline, intervention, washout, and crossover phases over an 12-week period.

Participants:

An a priori power analysis (G*Power) indicated that 19 participants are needed to detect a large effect (Cohen's d = 0.80, α = 0.05, power = 0.90). To allow for some expected attrition (~20%), 24 participants will be recruited.

Inclusion criteria:

* Age 40-65 years, BMI 25-35 kg/m²
* Full permanent dentition to first molar
* No diagnosed underbite, braces, dentures, or planned dental work
* Not currently using a CPAP device

Procedures:

Participants meeting inclusion criteria will undergo digital oral scans (upper, lower, and occlusal) to fabricate two custom devices. All scans will be completed at Tuscany Dental Centre (11300 Tuscany Blvd NW, Suite 2078, Calgary, AB T3L 2V7) and will be performed or overseen by Dr. Cam Brauer, a licensed dentist. The iTero digital oral scanner is a non-invasive, radiation-free optical imaging device used to obtain high-resolution 3D models of a participant's teeth and oral structures. The procedure involves using a handheld scanning wand to capture sequential images of the upper and lower arches and a brief bite registration. The wand does not contact any tissues, and the scan typically takes 8-12 minutes. This procedure is widely used in clinical practice and carries minimal risk. Potential minor discomforts may include mild jaw fatigue or a brief gag reflex, but no anesthetic or radiation is involved. All scan data are securely stored, de-identified, and transmitted in accordance with the study's data-management plan and relevant privacy regulations. Scans are performed by trained dental professionals following standard infection-control procedures.

The Placebo Device (PD) is a splint in centric occlusion with no mandibular advancement. The PX3™ Device advances the mandible 50-70% of maximum protrusion to improve alignment.

Each participant will receive a wrist-worn Garmin Forerunner 245 wearable device to continuously record sleep, HRV, and SpO2, except during bathing or charging. The device will be paired to the participant's smartphone using a study-specific Garmin Connect account created by the research team that does not contain personally identifying information. Data will be synced to the smartphone and retrieved by the research team on a rolling basis. Although the device is capable of collecting GPS data, GPS information will not be accessed, downloaded, or analyzed. Only sleep, HRV, and SpO2 metrics will be retained for research purposes. Data collection will occur over an 12-week period consisting of several phases: a 4-week baseline phase during which participants wear the monitor without any oral device; Phase 1 (3 weeks), where participants are randomized to either the PX3™ or placebo device; a 1-week washout period with no device use; Phase 2 (3 weeks), during which participants switch to the alternate device; and finally, a 1-week follow-up period of continued monitoring after completing both conditions.

Participants will wear the assigned oral appliance during sleep (mandatory) and may optionally use it during daytime. At each in-person visit, they will return devices and complete a survey on comfort, adherence, and perceived effects.

Participants will also maintain a nightly sleep log documenting their subjective sleep quality and any atypical factors that could influence restfulness (e.g., alcohol consumption, excessive exercise, illness, or travel). These notes will help contextualize variations in wearable-derived sleep and recovery metrics.

Data Analysis:

Sleep stage proportions (deep, light, REM, awake), HRV, and SpO2 data will be extracted from the wearable device for baseline and intervention phases. The percentage change in each variable will be calculated as:

% Change = [(Intervention - Baseline) / Baseline] × 100%

Paired t-tests will compare mean percentage changes between PX3™ and placebo conditions for sleep, HRV, and SpO2 outcomes. Statistical significance will be set at α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 40-65 years
* Male or female
* Body mass index (BMI) between 25 and 35 kg/m²
* Full set of permanent teeth to the first molar
* No clinically diagnosed underbite (Class III malocclusion)
* Generally healthy with no diagnosed sleep disorders
* Not currently using continuous positive airway pressure (CPAP) therapy
* Employed in predominantly desk-based or professional roles

Exclusion Criteria:

* Diagnosed underbite (Class III malocclusion)
* Current orthodontic treatment, braces, dentures, or pending dental work
* Use of CPAP therapy or diagnosis of severe sleep apnea
* Significant temporomandibular joint (TMJ) pain or dysfunction
* Current smoker or use of tobacco or vaping products
* Presence of major medical or psychiatric conditions that may affect sleep or autonomic function (e.g., cardiovascular disease, uncontrolled hypertension, anxiety, or depression)
* Pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Duration | Baseline (no oral appliance) and throughout each intervention phase while wearing the PX3™ device and the placebo device, through study completion (up to approximately 12 weeks)
  Total sleep duration will be measured using a wrist-worn Garmin Forerunner 245 wearable device. Sleep duration will be calculated as the total time classified as sleep during each recorded night across baseline and intervention phases.
  Unit of Measure:
  Minutes (or hours)
Sleep Stage Proportions | Baseline (no oral appliance) and throughout each intervention phase while wearing the PX3™ device and the placebo device, through study completion (up to approximately 12 weeks)
  Sleep stage proportions (deep sleep, light sleep, REM sleep, and awake time) will be measured using a wrist-worn Garmin Forerunner 245 wearable device. Sleep stage data will be recorded continuously during baseline and intervention phases and summarized as the proportion of total sleep time spent in each sleep stage.
  Unit of Measure:
  Percentage (%) of total sleep time
Heart Rate Variability (HRV) | Baseline (no oral appliance) and throughout each intervention phase while wearing the PX3™ device and the placebo device, through study completion (up to approximately 12 weeks)
  Heart rate variability will be measured using a wrist-worn Garmin Forerunner 245 wearable device. HRV data will be collected continuously during baseline and intervention phases and extracted for analysis using device-derived metrics.
  Unit of Measure:
  Milliseconds (ms)
Blood Oxygen Saturation (SpO2) | Baseline (no oral appliance) and throughout each intervention phase while wearing the PX3™ device and the placebo device, through study completion (up to approximately 12 weeks)
  Blood oxygen saturation (SpO₂) will be measured using a wrist-worn Garmin Forerunner 245 wearable device. SpO₂ data will be recorded during sleep periods throughout baseline and intervention phases and extracted for analysis.
  Unit of Measure:
  Percentage (%)

SECONDARY OUTCOMES:
Participant Comfort With the Device | Baseline (no oral appliance) and throughout each intervention phase while wearing the PX3™ device and the placebo device, through study completion (up to approximately 12 weeks)
  Participant-reported comfort while wearing the device will be assessed using a survey administered after each study condition.
  Unit of Measure:
  Likert scale (as defined in the survey)
Participant Adherence to Device Use | Immediately after each intervention phase (after Condition 1 and after Condition 2)
  Participant adherence to wearing the device as instructed will be assessed using a self-reported survey administered after each study condition.
  Unit of Measure:
  Likert scale or percentage of prescribed wear time (as defined in the survey)
Participant Experience Using the Device | Immediately after each intervention phase (after Condition 1 and after Condition 2)
  Overall participant experience using the device will be assessed using a survey administered after each study condition.
  Unit of Measure:
  Likert scale (as defined in the survey)
Participant-Perceived Effects of the Device | Immediately after each intervention phase (after Condition 1 and after Condition 2)
  Participant-perceived effects of the device on sleep, recovery, or daily functioning will be assessed using a survey administered after each study condition.
  Unit of Measure:
  Likert scale (as defined in the survey)

CONTACTS AND LOCATIONS:
Overall Officials: Christian A Clermont, PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Data collected in this study include detailed physiological and health-related measures, and sharing individual-level data could increase the risk of participant re-identification. Only aggregated, de-identified summary results will be reported and shared in publications or presentations, in accordance with institutional ethics approval and data-governance policies.